CLINICAL TRIAL: NCT02505841
Title: Transversus Abdominis Plane (TAP) Block for Laparoscopic Appendicectomy in Children: Opioid Saving and Alternative in the Curarization
Brief Title: Transversus Abdominis Plane Block for Laparoscopic Appendicectomy in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9488; 2014-A01431-46 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-06-22; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-05

CONDITIONS: Laparoscopic Appendectomy
Keywords: Appendectomy; Laparoscopy; pediatric surgery
MeSH Terms: interventions — Ropivacaine; Dental Occlusion; Curare; Succinylcholine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Curare: Atracurium injection at 0.5 mg/kg
  Interventions: Drug: Curare
- Group 2 (Experimental): TAP block and curare: Ultrasound-guided transversus abdominis plane block wih Ropivacaine injection 0.2% at 0.3 ml/kg then atracurium injection at 0.5 mg/kg
  Interventions: Other: TAP block with Ropivacaine; Drug: Curare
- Group 3 (Experimental): TAP block: Ultrasound-guided transversus abdominis plane block wih Ropivacaine injection 0.2% at 0.3 ml/kg
  Interventions: Other: TAP block with Ropivacaine

INTERVENTIONS:
Other: TAP block with Ropivacaine — Ultrasound-guided transversus abdominis plane block wih Ropivacaine injection 0.2% at 0.3 ml/kg
  Other Names: Transversus abdominis plane (TAP) block with ropivacaine
  Arms: Group 2; Group 3
Drug: Curare — Atracurium injection at 0.5 mg/kg at least 3 minutes before the surgical incision
  Other Names: Succinylcholine
  Arms: Group 1; Group 2

SUMMARY:
The transversus abdominis plane (TAP) block is a regional anesthetic technique for post operative pain control after abdominal surgical procedures. Its effectiveness in children undergoing laparoscopic appendectomy has not been demonstrated. The investigators evaluate its analgesic efficacy over the first 24 post operative hours.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in surgery and infantile anesthesia unit or admitted in emergencies for an laparoscopic appendectomy surgery.
* Patient whose general state corresponds to the classification of the American Society of Anesthesiologists (ASA) I to II
* Patient member in a national insurance scheme

Exclusion Criteria:

* Patient with drilled appendicitis or peritonitis
* Patient with a contraindication to local anesthesics
* Patient with a contraindication to TAP block
* Patient with allergies or known hypersensitivity to curare

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Painkiller of help consumption | up to 24 hours after surgery
  Quantity of analgesic of help (Nalbuphine, Nubain®, Dupont Pharma, Paris, France) taken after the surgery.

SECONDARY OUTCOMES:
Pain intensity after surgery | up to 24 hours
  The post-operative pain will be estimated from the arrival in recovery room with the Face Legs Activity Cry Consolability (FLACC) scale.
First demand of analgesic of help | up to 12 hours
  First demand of analgesic of help (Nubain ®) after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maud MM Maniora, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- CHRU Montpellier, Montpellier, France